CLINICAL TRIAL: NCT05785065
Title: Randomized Double-Blind Placebo-Controlled Clinical Trial to Assess the Efficacy of Mycophenolate Mofetil in Subclinical Interstitial Lung Disease Associated With Systemic Sclerosis: a Feasibility Study
Brief Title: Mycophenolate Mofetil in Systemic Sclerosis With Subclinical Interstitial Lung Disease
Acronym: SSc-mILD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: McGill University (Other); University of Calgary (Other); Jewish General Hospital (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Sclérodermie Québec (Unknown); Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MP-02-2023-11180
Record Dates: First submitted 2023-02-07; First posted 2023-03-27 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Systemic Sclerosis With Lung Involvement; Systemic Sclerosis; Interstitial Lung Disease
Keywords: Systemic sclerosis; Mycophenolate mofetil; Interstitial lung disease
MeSH Terms: conditions — Scleroderma, Systemic; Lung Diseases, Interstitial | interventions — Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to treatment group or placebo group in a 1:1 ratio and stratified according to the presence of anti-topoisomerase I autoantibody.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant, the physician, the study investigators and the research personnel will be blinded to treatment allocation, whereas the dispensing pharmacy will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mycophenolate mofetil (Experimental): 2 to 4 capsules of mycophenolate mofetil twice daily.
  Interventions: Drug: Mycophenolate Mofetil
- Placebo (Placebo Comparator): 2 to 4 capsules of placebo twice daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mycophenolate Mofetil — The participant will receive 500 mg to 1000 mg twice daily of mycophenolate mofetil administered orally for 96 weeks.
  The dose scheduling will be as follow:
  Weeks 1 and 2: 500 mg twice a day Weeks 3 and 4: 750 mg twice a day Weeks 5 to 96: 1000 mg twice a day
  Arms: Mycophenolate mofetil
Other: Placebo — The participant will receive 500 mg to 1000 mg twice daily of placebo administered orally for 96 weeks.
  The dose scheduling will be as follow:
  Weeks 1 and 2: 500 mg twice a day Weeks 3 and 4: 750 mg twice a day Weeks 5 to 96: 1000 mg twice a day
  Arms: Placebo

SUMMARY:
The goal of this pilot study is to assess the feasibility of a larger study on the efficacy of mycophenolate mofetil in people diagnosed with systemic sclerosis with mild lung involvement. Participants will be recruited over 12 months at 3 academic centers and assigned randomly to receive either mycophenolate mofetil or placebo, a look-alike substance that contains no active drug, for 96 weeks.

DETAILED DESCRIPTION:
Background: Systemic sclerosis (SSc, scleroderma) is a rare but life-threatening systemic autoimmune disease characterized by microvasculopathy, serum autoantibodies, inflammation and fibrosis of the skin and internal organs. Early rapidly progressive SSc remains the most lethal autoimmune rheumatic disease, with over 60% mortality at 5 years in high-risk patients. Interstitial lung disease (ILD) is the leading cause of SSc-related mortality and affects over half of SSc patients. SSc-ILD is currently treated with immunosuppressive and anti-fibrotic drugs, with the first-line treatment being mycophenolate mofetil (MMF), although treatments have modest benefits when initiated in advanced stages of disease. Emerging data suggest that earlier treatment, when lung function is still normal despite evidence of ILD on computed tomography scan ("subclinical SSc-ILD"), may lead to improved outcomes, suggesting a window of treatment opportunity.

Research Aims: The goal of the proposed pilot RCT is to establish the feasibility of a phase III RCT that will assess the efficacy of MMF in subclinical SSc-ILD. Specifically, we aim to:

1. Determine the rate of patient recruitment at three centers over one year, and identify barriers and solutions to recruitment;
2. Determine the proportion of participants receiving the allocated treatment and with complete primary efficacy outcome data at 48 and 96 weeks; and
3. Generate preliminary data on clinical efficacy outcomes that will contribute information to the analysis of the phase III trial through a Bayesian inference framework.

Methods: Participants will be adults with SSc, ILD diagnosed within the past 3 years and a normal forced vital capacity (≥ 80%). Participants will be recruited over 12 months at 3 academic centers affiliated to the Canadian Scleroderma Research Group. Eligible participants will be assigned using stratified randomization to receive either MMF (up to 2 grams daily) or placebo for 96 weeks. The primary feasibility outcome will be the rate of recruitment per site over 12 months. A Bayesian approach will be used to estimate the probability of reaching the target sample size based on observed recruitment rates, with decision rules to continue, adapt, or stop the trial. Data collected on the primary clinical efficacy outcome (annual rate of decline in forced vital capacity over 96 weeks) will be used to inform the analysis of the phase III trial (as an informative prior) through a Bayesian inference framework.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent and adhere to study protocol;
2. Women and men of all race/ethnicity, aged 18 years and older;
3. SSc based on 2013 ACR-EULAR classification criteria;
4. Presence of interstitial lung disease on HRCT scan, obtained within 12 months before screening, that shows fibrosis affecting less than 20% of the lungs, as confirmed by an expert radiologist;
5. Diagnosis of ILD within 7 years before screening;
6. Forced vital capacity of 80% predicted and above, on pulmonary function tests obtained within 6 months before screening;
7. Able to communicate in French or English;

Exclusion Criteria:

1. Progressive pulmonary fibrosis, defined as at least two of three criteria (worsening symptoms, radiological progression, and physiological progression) occurring within the past year with no alternative explanation, as defined by the 2022 ATS/ERS/JRS/ALAT Clinical Practice Guideline;
2. Use of medications with putative lung disease-modifying properties:

   1. Current use of MMF, mycophenolic acid, azathioprine, calcineurin inhibitors (e.g. tacrolimus, cyclosporin A), tocilizumab, nintedanib, pirfenidone or corticosteroids (Prednisone equivalent dose >10 mg/day) at time of screening
   2. Cyclophosphamide within one year prior to screening
   3. Rituximab within 6 months prior to screening
   4. Cell therapies (including stem cell transplantation) within one year prior to screening
3. Current use of other biological, targeted synthetic or investigational products with immunosuppressive effects (e.g. TNF inhibitors, abatacept, tofacitinib) at time of screening
4. Any contraindication to MMF, including:

   1. Pregnancy and/or breastfeeding
   2. Female of childbearing potential not using reliable method of contraception
   3. Persistent leucopenia (white blood cell count <3.0 x103/μL)
   4. Persistent thrombocytopenia (platelet count <100 x103/μL)
   5. Persistent anemia (hemoglobin <100 g/L)
   6. Baseline liver enzymes (alanine transaminase (ALT) or aspartate transaminase (AST)) or bilirubin >1.5 times the upper limit of normal, other than due to Gilbert's disease
   7. Uncontrolled congestive heart failure
   8. Active infection (lung or elsewhere)
   9. Active solid or hematological malignancy (other than basal cell cancer of the skin or cervical carcinoma in situ removed entirely by biopsy)
   10. Active peptic ulcer disease
   11. Other serious concomitant medical illness, unreliability or drug abuse that might compromise the patient's ability to safely take MMF
   12. Use of drugs or products with significant interactions with MMF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Total number of potentially eligible patients identified per site | Over one year
Proportion of potentially eligible patients who provide consent per site | Over one year
Proportion of consented participants who meet the eligibility criteria per site | Over one year
Monthly rate of randomized participants per site | Over one year
Adherence to treatment as assessed by Participant Dosing Diaries | From the first dose to the last dose taken for each participant, up to 96 weeks
Drug adherence rate as assessed by Pharmacy Accountability Logs | From the first dose to the last dose taken for each participant, up to 96 weeks
Adherence to the study protocol as assessed by the number of protocol deviations | Over total study period (up to 96 weeks per participant)
Proportion of participants intolerant to the study drug who discontinue trial treatment | Over total study period (up to 96 weeks per participant)
Proportion of participants receiving the allocated treatment at 48 weeks | At 48 weeks
Proportion of participants receiving the allocated treatment at 96 weeks | At 96 weeks
Proportion of participants with complete primary efficacy outcome data at 48 weeks | At 48 weeks
Proportion of participants with complete primary efficacy outcome data at 96 weeks | At 96 weeks
Proportion of participants lost to follow-up | Over total study period (up to 96 weeks per participant)

SECONDARY OUTCOMES:
Frequency of treatment-related adverse events | Over total study period (up to 96 weeks per participant)
  Incidence and severity of AEs, with severity determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)

OTHER OUTCOMES:
Annual rate of decline in percent (%) predicted forced vital capacity (FVC) over 48 weeks | Over 48 weeks
Annual rate of decline in percent (%) predicted forced vital capacity (FVC) over 96 weeks | Over 96 weeks
Proportion of participants having clinically meaningful progression | Over total study period (up to 96 weeks per participant)
  Clinically meaningful progression defined by the Outcome Measures in Rheumatology (OMERACT) for connective tissue disease-associated interstitial lung diseases (CTD-ILD) (defined as a ≥10% relative decline in FVC from baseline, or a ≥5% to <10% relative decline in FVC associated with a ≥15% relative decline in diffusion capacity [DLCO])
Time to clinically meaningful progression | Over total study period (up to 96 weeks per participant)
  Clinically meaningful progression as defined by Outcome Measures in Rheumatology (OMERACT) for connective tissue disease- associated interstitial lung diseases (CTD-ILD) (defined as a ≥10% relative decline in FVC from baseline, or a ≥5% to <10% relative decline in FVC associated with a ≥15% relative decline in diffusion capacity [DLCO])
Proportion of participants having an absolute decrease in FVC of at least 3.3% predicted | Over total study period (up to 96 weeks per participant)
  An absolute decrease in FVC of at least 3.3% predicted was proposed as the minimal clinically important difference estimate for worsening of FVC in patients with SSc-ILD.
Time to an absolute decrease in FVC of at least 3.3% predicted | Over total study period (up to 96 weeks per participant)
  An absolute decrease in FVC of at least 3.3% predicted was proposed as the minimal clinically important difference estimate for worsening of FVC in patients with SSc-ILD.
Proportion of participants having progressive pulmonary fibrosis | Over total study period (up to 96 weeks per participant)
  Progressive pulmonary fibrosis defined by 2022 ATS/ERS/JRS/ALAT guidelines
Time to progressive pulmonary fibrosis | Over total study period (up to 96 weeks per participant)
  Progressive pulmonary fibrosis defined by 2022 ATS/ERS/JRS/ALAT guidelines
Annual rate of decline in percent (%) predicted total lung capacity over 48 weeks | Over 48 weeks
Annual rate of decline in percent (%) predicted total lung capacity over 96 weeks | Over 96 weeks
Annual rate of decline in percent (%) predicted diffusion capacity for carbon monoxide (DLCO) over 48 weeks | Over 48 weeks
Annual rate of decline in percent (%) predicted DLCO over 96 weeks | Over 96 weeks
Change from baseline in percent (%) extent of ILD, ground-glass opacities, reticular infiltrates and honeycombing, and in pulmonary vessel volume at 48 weeks | At 48 weeks
  Measured on high-resolution computed tomography chest scan using automated lung texture analysis
Change from baseline in percent (%) extent of ILD, ground-glass opacities, reticular infiltrates and honeycombing, and in pulmonary vessel volume at 96 weeks | At 96 weeks
  Measured on high-resolution computed tomography chest scan using automated lung texture analysis
Change from baseline in St-George Respiratory Questionnaire at 48 weeks | At 48 weeks
  Scores range from 0 to 100, with higher scores indicating more limitations.
Change from baseline in St-George Respiratory Questionnaire at 96 weeks | At 96 weeks
  Scores range from 0 to 100, with higher scores indicating more limitations.
Change from baseline in Leicester Cough Questionnaire at 48 weeks | At 48 weeks
  Scores (total) range from 3 to 21, with higher scores indicating less limitations.
Change from baseline in Leicester Cough Questionnaire at 96 weeks | At 96 weeks
  Scores (total) range from 3 to 21, with higher scores indicating less limitations.
Change from baseline in health assessment questionnaire modified for scleroderma at 48 weeks | At 48 weeks
  The SHAQ consists of the Health assessment questionnaire (HAQ) and visual analogue scales for pain, patient global assessment, vascular, digital ulcers, lung involvement and gastrointestinal involvement. Scores range from 0 to 3, with higher scores indicating more limitations.
Change from baseline in health assessment questionnaire modified for scleroderma at 96 weeks | At 96 weeks
  The SHAQ consists of the Health assessment questionnaire (HAQ) and visual analogue scales for pain, patient global assessment, vascular, digital ulcers, lung involvement and gastrointestinal involvement. Scores range from 0 to 3, with higher scores indicating more limitations.
Change from baseline in 36-items short form survey (SF-36) at 48 weeks | At 48 weeks
  Eight scales with scores range from 0 to 100, with higher scores indicating less limitations.
Change from baseline in 36-items short form survey (SF-36) at 96 weeks | At 96 weeks
  Eight scales with scores ranging from 0 to 100, with higher scores indicating less limitations.
Change from baseline in EuroQoL five dimensions (EQ-5D-5L) at 48 weeks | At 48 weeks
  The EQ-5D-5L questionnaire possesses 5 levels for each of the five dimensions. The five dimensions are mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with the following possible five responses: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Scores are converted into an index value ranging from 0 to 1, with higher scores indicating better health state.
Change from baseline in EuroQoL five dimensions (EQ-5D-5L) at 96 weeks | At 96 weeks
  The EQ-5D-5L questionnaire possesses 5 levels for each of the five dimensions. The five dimensions are mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with the following possible five responses: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. Scores are converted into an index value ranging from 0 to 1, with higher scores indicating better health state.
Change from baseline in patient global assessment at 48 weeks | At 48 weeks
  Visual analogue scale from 0 to 10, with higher scores indicating worse disease.
Change from baseline in patient global assessment at 96 weeks | At 96 weeks
  Visual analogue scale from 0 to 10, with higher scores indicating worse disease.
Change from baseline in physician global assessment at 48 weeks | At 48 weeks
  Visual analogue scale from 0 to 10, with higher scores indicating worse disease.
Change from baseline in physician global assessment at 96 weeks | At 96 weeks
  Visual analogue scale from 0 to 10, with higher scores indicating worse disease.
Change from baseline in 6-minute walk oxygen saturation at 48 weeks | At 48 weeks
  Oxygen saturation at nadir during the 6-minute walk test
Change from baseline in 6-minute walk oxygen desaturation at 96 weeks | At 96 weeks
  Oxygen saturation at nadir during the 6-minute walk test
Change from baseline in modified Rodnan skin score (mRSS) at 48 weeks | At 48 weeks
  Scores range from 0 to 51, with higher scores indicating more skin involvement.
Change from baseline in modified Rodnan skin score (mRSS) at 96 weeks | At 96 weeks
  Scores range from 0 to 51, with higher scores indicating more skin involvement.
Change from baseline in nailfold capillary density at 48 weeks | At 48 weeks
  Mean number of capillaries per mm
Change from baseline in nailfold capillary density at 96 weeks | At 96 weeks
  Mean number of capillaries per mm
Change from baseline in nailfold capillaroscopy abnormalities and patterns at 48 weeks | At 48 weeks
  Ectasias/megacapillaries are scored using a semi-quantitative scale (0 = no, 1 = ≤33%, 2= 33-66%, and 3 = ≥66% abnormalities/linear mm)
Change from baseline in nailfold capillaroscopy abnormalities and patterns at 96 weeks | At 96 weeks
  Ectasias/megacapillaries are scored using a semi-quantitative scale (0 = no, 1 = ≤33%, 2= 33-66%, and 3 = ≥66% abnormalities/linear mm)
Change from baseline in quantitative SSc autoantibody titers at 48 weeks | At 48 weeks
Change from baseline in quantitative SSc autoantibody titers at 96 weeks | At 96 weeks
Change from baseline in Krebs von Lungen 6 (KL-6) titers at 48 weeks | At 48 weeks
Change from baseline in Krebs von Lungen 6 (KL-6) titers at 96 weeks | At 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Hoa, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (3):
- Canada (3):
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital - CIUSSS-COMTL, Montreal, Quebec
  - Institut Universitaire de Cardiologie et Pneumologie de Québec, Québec, Quebec